CLINICAL TRIAL: NCT04032795
Title: Evaluation of Efficacy of Lycium Barbarum Polysaccharide in People With Subthreshold Depression: a Randomized, Placebo-controlled Trial
Brief Title: Evaluation of Efficacy of Lycium Barbarum Polysaccharide in People With Subthreshold Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Collaborators: Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Kangguang Lin, Deputy director, Department of Affective disorders, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Guangzhou Brain LBP
Record Dates: First submitted 2019-07-19; First posted 2019-07-25 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Subthreshold Depression; Depressive Symptoms; Anxious Symptoms
Keywords: Major Depressive Disorder; Lycium barbarum polysaccharide; depressive symptoms; anxious symptoms
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — lycium barbarum polysaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lycium barbarum polysaccharide (LBP) (Experimental): Experimental group takes LBP tablet (300mg/day) for 6 weeks
  Interventions: Dietary Supplement: Lycium barbarum polysaccharide
- Placebo (Placebo Comparator): Placebo control group takes placebo 6 weeks. The placebos are the same with the LBP tablets in appearance and taste.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lycium barbarum polysaccharide — Experimental group takes Lycium barbarum polysaccharide (LBP) tablet (300mg/day)for 6 weeks
  Arms: Lycium barbarum polysaccharide (LBP)
Dietary Supplement: Placebo — Placebo-controlled group take he placebo capsules that are identical in shape, color, and taste to LBP tablet.
  Arms: Placebo

SUMMARY:
Lycium barbarum, a traditional Chinese herbal medicine, is a commonly used herb in the traditional Chinese pharmacopoeia . Its main active ingredient, lycium barbarum polysaccharide (LBP), is reported to have neuroprotective effects. Animal studies suggested that LBP has neuroprotective effect on optic ganglion cells. In animal models of depression, LBP can improve depressive symptom by improving synaptic plasticity. However, its clinical effect remains to be studied. We will conduct a 6-week double-blind, randomized, placebo-con-trolled trial in people with subthreshold depression.The purpose of this clinical trial is to investigate the efficacy of LBP in people with subthreshold depression.

ELIGIBILITY:
Inclusion Criteria:

1. 15-25 scores in the Beck Depression Rating Scale (BDI- II)
2. There is no contraindication of taking LBP.

Exclusion Criteria:

1. Current treatment for a mental health problem from a mental health professional
2. Current and lifetime history of psychiatric disorders (e.g major depressive disorder, as ascertained by CIDI
3. Systemic disease requiring regular medication.
4. There are suicidal ideation, suicidal attempt, suicide behavior and attempted suicide.
5. Dislike of or allergy to goji berry
6. Hormone or Endocrine therapeutic drugs are being taken.
7. Long-term use of lycium chinensis in recent three months

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean changes from baseline in the 21-item Hamilton Depression Rating Scale (24-HAMD) | 6 weeks
  The 24-item HAM-D scale is widely used to assess the severity of depression.The scale is a 21-item assessment used to measure depression severity. Items were rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score ranging from 0 (not at all depressed) to 64 (severely depressed).

SECONDARY OUTCOMES:
Changes in The Screen for Child Anxiety Related Disorders (SCARED) | 4 and 6 weeks
  The SCARED is a child and parent self-report instrument used to screen for childhood anxiety disorders including general anxiety disorder, separation anxiety disorder, panic disorder, and social phobia.
Changes in sleep quality | 6 weeks
  Changes in Pittsburgh Sleep Quality Index (PSQI)
Depression severity as measured by BDI2 and Kessler Scale (K10) | 6 weeks
  The Kessler psychological distress scale (K10) is a widely used, simple self-report measure of psychological distress which can be used to identify those in need of further assessment for anxiety and depression.
Mean change from baseline in the Beck Depression Inventory-II (BDI-2)total scores | 6 week
  The BDI-II is a 21-item self-report measure of depressive symptom.Remission was defined as equal or less than 8 scores on BDI-2.

OTHER OUTCOMES:
Treatment-emergent symptom side effect (TESS) scale. | 4 and 6 weeks
  Side effect was evaluated by treatment-emergent symptom side effect (TESS) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kwok-Fai So, PhD, Study Chair — Guangzhou Medical University; Kangguang Lin, MD,PhD, Study Director — Guangzhou Brain Hospital (Guangzhou Huiai Hospital);The fifth affiliated hospital of Guangzhou Medical University; Xuan Mo, MD, Principal Investigator — Fifth Affiliated Hospital of Guangzhou Medical University; Guiyun Xu, MD, Principal Investigator — Guangzhou Brain Hospital (Guangzhou Huiai Hospital)
Locations (1):
- The Affiliated Fifth Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li X, Mo X, Liu T, Shao R, Teopiz K, McIntyre RS, So KF, Lin K. Efficacy of Lycium barbarum polysaccharide in adolescents with subthreshold depression: interim analysis of a randomized controlled study. Neural Regen Res. 2022 Jul;17(7):1582-1587. doi: 10.4103/1673-5374.330618. PMID 34916444